# Therapeutic Effect Of Luteolin Natural Extract Versus Its Nanoparticles On Tongue Squamous Cell Carcinoma Cell Line: In Vitro Study

**September**, 18 2017

# **Presented by:**

Safaa Mohamed Ibrahim Baz

# **List of Contents:**

| Administrative Information | 4 |
|-------------------------------------------|----|
| 1. Title | 4 |
| 2. Protocol Version | 4 |
| 3. Roles and Responsibilities | 4 |
| Steering Committees | 4 |
| Assessment and Auditing | 5 |
| Research Ethics Approval | 5 |
| Access to Data | 5 |
| Dissemination Policy | 5 |
| Funding | 5 |
| 1. Introduction | 6 |
| 1. 1. Background and Scientific Rationale | 6 |
| 1. 2. Objectives | 8 |
| 2. PICO | 9 |
| 3. Research Question | 9 |
| 4. Material and Methods | 9 |
| 4. 1. Collecting samples | 9 |
| 4. 2. Materials | 10 |
| 4. 3. Methods | 10 |
| 4. 4. Sample size | 13 |
| 4. 5. Randomization | 14 |
| 4. 6. Blinding and assessment | 14 |
| 4. 7. Statistical methodology | 14 |

| 5. | Results | 14 |
|----|----------------------------------------|----|
| | 5. 1. Outcome(s) (O) | 14 |
| | 5. 2. Testing the samples | 14 |
| 6. | Protocol amendments | 15 |
| 7. | Search strategy | 15 |
| | 7. 1. The PRISMA Statement | 15 |
| | 7. 2. Summary of finding tables (SOFT) | 24 |
| 8. | References | 29 |

### **Administrative Information:**

#### \* Title:

Therapeutic Effect of Luteolin Natural Extract Versus Its Nanoparticles on Tongue Squamous Cell Carcinoma Cell Line: In Vitro Study

### \* Protocol Version:

Version (1)

### \* Roles and Responsibilities:

#### 1-The Principle Supervisor:

➤ **Prof. Dr. Heba Ahmad Farag** (H.F.), Professor of Oral & Maxillofacial Pathology, Faculty of Oral & Dental Medicine, Cairo University.

#### 2-The Assistant Supervisor:

➤ Dr. Safa Fathy Abd-Elghany (S.F.), Assistant Professor of Oral & Maxillofacial Pathology, Faculty of Oral & Dental Medicine, Cairo University.

#### **3-The Investigators:**

- ➤ **Dr. Esam Rashwan** (E.R.), Assistant Professor and Head of Confirmatory Diagnostic Unit, VACSERA-Egypt
- Safaa Mohamed Mohamed Ibrahim Baz (S.B.), (The Principle Investigator)
  Assistant Lecturer of Oral & Maxillofacial Pathology, Faculty of Oral & Dental
  Medicine, BUE.

## **Steering Committees:**

- 1. Oral & Maxillofacial Pathology Department Board, Faculty of Dentistry, Cairo University.
- 2. Evidence Based Committee, Faculty of Dentistry, Cairo University.

- 3. Ethics Committee, Faculty of Dentistry, Cairo University.
- 4. Higher Education and Research Committee.
- 5. Faculty Board.

## **Assessment and Auditing:**

#### The assessment and auditing of the study design was done by:

- 1. Oral & Maxillofacial Pathology Department Board, Faculty of Dentistry, Cairo University.
- 2. Evidence Based Committee, Faculty of Dentistry, Cairo University.

## **Research Ethics Approval:**

This protocol will be reviewed by:

Ethical Committee, Faculty of Dentistry, Cairo University.

## **Access to Data:**

All Investigators of the study will be given access to the data.

## **Dissemination Policy:**

Study results will be published as a partial fulfillment of the requirements for the PhD degree in Oral & Maxillofacial Pathology.

## **Funding:**

Self-funding.

## 1. Introduction:

### 1. 1. Background and Scientific Rationale:

Cancer still one of the most lethal diseases causing an expansive number of deaths globally. In 2015, the WHO stated that the number of individuals died from cancer all over the world was about 8.8 million and indicated that by 2030 this number will show a marked elevation exceeding 13 million <sup>1</sup>. Among malignancies, oral cancer is the sixth most common neoplasm around the world. Oral squamous cell carcinoma (OSCC) is the most widely recognized oral malignancy representing almost 90% of the oral cancers worldwide <sup>2</sup>, with a variable global incidence which differs in each area according to the exposure to specific risk factors <sup>3</sup>.

For treatment of OSCC, the primary therapeutic modalities are surgical intervention, radiotherapy, and chemotherapy <sup>4,5</sup>. Chemotherapeutic agents play a vital role in the treatment of malignancy by killing cancerous cells. Nevertheless, they cause cytotoxic impacts to the adjacent normal cells and leave behind tissue resistance which is considered to be serious obstructions encountered the chemotherapy treatment. Therefore, the scientific community has the responsibility to discover an alternative naturally occurring drug with minimal side effects and maximal efficacy in cancer therapy <sup>6</sup>.

plant-derived compounds, flavonoids accepted natural chemotherapeutic agents 7 with many points of interest over the traditional chemotherapy, (e.g. better bioavailability, lower toxicological profile, as well as affordability) 8. Luteolin, 3',4',5,7-tetrahydroxyflavone, is a naturally occurring flavonoid isolated from a wide variety of medicinal herbs, fruits, and vegetables (e.g. parsley, artichoke, celery, onion leaves, broccoli, carrots, green and sweet bell pepper, perilla leaves and chrysanthemum flowers) 9-<sup>12</sup>. Luteolin has been appeared to display several significant biological properties, ranging from antioxidant and anti-inflammatory effects chemoto cancer therapeutic/chemoprevention activities <sup>13</sup>.

A recent in vitro and in vivo study has demonstrated that luteolin and its nanoparticles have anticancer activity against cells of lung cancer and squamous cell carcinoma of head and neck <sup>14</sup>.

Regarding the therapeutic effect of luteolin, a study on hepatic carcinoma cells has revealed a high level of apoptotic cells (reached to  $58.18\pm2.11\%$ ) after 50  $\mu$ M luteolin treatment for 24 hours  $^{15}$ .

To provide a magnificent enhancement in the treatment effectiveness and overcome the undesired current cancer therapy toxicity, the researchers have potentially turned to nanotechnology-based regimens incorporation with several promising qualities over the conventional chemotherapy <sup>16</sup>. Furthermore, the anticancer activity of nano-luteolin (nanoparticle delivery of luteolin) has suggested many advantages superior to luteolin and may have potential application in clinical settings <sup>17</sup>.

## 1. 2. Objectives:

In vitro study to examine whether luteolin and nano-luteolin exert an inhibitory effect on tongue squamous cell carcinoma cell line by inducing apoptosis, and to assess if nano-luteolin has more efficient apoptotic activity than luteolin on tongue squamous cell carcinoma cell line.

### **2. PICO:**

**Population (P):** Cultured tongue squamous cell carcinoma cell line.

#### **Intervention (I):**

> I 1: Application of luteolin

> I 2: Application of nano-luteolin

**Control (C):** No treatment.

#### Outcome(s) (O):

**Primary O:** Apoptosis (Gene expression of Caspase 3).

> Secondary O: Cytotoxicity/Cell viability.

| Outcome | Outcome name | Measuring Device | Measuring Unit |
|---|---|---|---|
| Primary | Apoptosis (Gene expression of Caspase 3) | RT-qPCR system <sup>18</sup> . | fold-changes |
| Secondary | Cytotoxicity/Cell viability | MTT assay using an ELISA<br>Reader <sup>19</sup> . | Micromolar (μM) |

#### Study design:

In vitro study

## 3. Research Question:

Do luteolin and nano-luteolin natural extracts exert an inhibitory effect on tongue squamous cell carcinoma cell lines by inducing apoptosis? Is nano-luteolin more efficient than luteolin in inducing apoptosis on tongue squamous cell carcinoma cell line?

## 4. Material and Methods:

## 4. 1. Collecting samples:

Tongue squamous cell carcinoma cell line will be purchased from veterinary serum & vaccine research institute (VACSERA), supplied with compatible nutrient media.

### 4. 2. Materials:

### **4. 2. 1. Intervention (I):**

- 1. Luteolin (Sigma-Aldrich)
- 2. Nano-luteolin (Luteolin nanoparticles prepared using ultrasonication nanotechnology)

### 4. 2. 2. Check list for the used drug:

| Item | Description |
|---|---|
| Name, common names and family name | Luteolin, 3',4',5,7-Tetrahydroxyflavone; Flavones, Flavonoids |
| Used product | Luteolin (Sigma-Aldrich) |
| Form | Powder |
| Color | Yellow |
| The type and concentration of solvent used | Ethanol (4.90 - 5.10 mg/ml) |
| Nano-luteolin | Luteolin nanoparticles prepared using ultrasonication nanotechnology |

## 4. 3. Methods:

All the steps of the current experiment will take place in Confirmatory Diagnostic Unit, R and D sector, VACSERA-Egypt, by E.R. and S.B.

### 4. 3. 1. Sample preparation: (According to ATCC\* protocol)

#### [Continuous Cell Line Cell Culture Protocol]

#### 1. Examination:

E.R. and S.B. will examine the culture prior to subcultivation using an inverted phase contrast microscope, and will check the general appearance of the culture.

#### 2. Cell harvesting:

When using 0.1% Trypsin solution for enzymatic dissociation:

- a) E.R. and S.B. will remove the old medium and discard it.
- b) We will rinse the cell monolayer gently.
- c) Then we will add the enzyme solution and incubate the culture until the cells are freleased.

#### 3. Cell counting:

To determine growth rates or set up cultures at known concentrations it is necessary to count the cell suspension.

- a) E.R. and S.B. will remove 0.5mL sample and place it in a tube for counting, with adding the vital stain Trypan blue. We will withdraw 20µL of the sample with a wide tip pipettor and carefully load a clean hemacytometer.
- b) We will count a viable cell count. We will calculate the number of viable cells/mL and the total cell number.

#### 4. Plating:

After making the appropriate dilutions, E.R. and S.B. will add the correct amount of cells to each culture vessel. Then we will add fresh medium to bring the cell culture vessel to its recommended working volume.

#### 5. Incubation:

- a) E.R. and S.B. will leave caps on flasks slightly loosened and place them on a shelf in a 37°C, humidified CO<sub>2</sub> incubator\*.
- b) We will examine culture daily and will change medium as needed.

<sup>\*</sup> Thermo Scientific Heraeus, UK.

#### 4. 3. 2. MTT assay: (According to Sigma-Aldrich protocol)

### [IC50 Calculation and MTT Assay with ELISA reader\* Protocol]

#### $\Rightarrow$ IC50 calculation:

- After plating and 24 hours incubation of the cell culture, E.R. and S.B. will remove the cell culture from incubator into laminar flow hood, and then apply to a 96-well plate (about 25,000-30,000 cells per well).
- E.R. and S.B. will add the drug with five serial concentrations (100, 10, 1, 0.1, and  $0.01 \mu g/mL$ ) to calculate the IC<sub>50</sub>% concentration in Micromolar ( $\mu M$ ).

#### $\Rightarrow$ MTT Assay should include:

- Blank wells containing medium only.
- Untreated control cells.
- Test cells treated with either luteolin or nano-luteolin with IC<sub>50</sub>% concentration.
  - 1) After plating and 24 hours incubation of the cell culture, E.R. and S.B. will remove the cell culture from incubator into laminar flow hood, and then apply to a 96-well plate (about 25,000-30,000 cells per well).
  - 2) E.R. and S.B. will reconstitute each vial of MTT to be used with 3 ml of medium or balanced salt solution without phenol red and serum. We will add the reconstituted MTT in an amount equal to 10% of the culture medium volume.
  - 3) We will return cultures to incubator for 2-4 hours until purple precipitate is visible.
  - 4) At the end of the incubation period, we will remove the cultures from incubator and dissolve the resulting purple formazan crystals by adding an amount of MTT Solubilization solution equal to the original culture medium volume.
  - 5) Well mixing will improve dissolution.
  - 6) We will measure absorbance spectrophotometrically at a wavelength of 450nm.

<sup>\*</sup> Bioline Technologies, India.

#### **4. 3. 3. RT-PCR:** (According to Bio-Rad Laboratories protocol)

### [One-step Rotor-Gene Q Real-Time PCR System\* Protocol]

1. Treatment of cell culture:

After plating and 24 hours incubation of the cell culture, E.R. and S.B. will treat the flask with the  $IC_{50}\%$  concentration of the drug for the treatment incubation time.

- 2. We will harvest cells, then lysis cells.
- 3. E.R. and S.B. will prepare all the required components (including SYBR® Green one-step kit, SYBR® Green Supermix, sequence-specific primers for Caspase, necessary enzymes and a buffer solution) except RNA on ice reaction set up.
- 4. We will mix the reaction set up thoroughly then dispense into the PCR tube.
- 5. Then we will add the template RNA to the PCR tube, seal and shake the tube.
- 6. The thermal cycling protocol will be programmed according to the steps which are summarized in the following table:

| The first cycle | The second cycle The next 35-40 cyc | | 35-40 cycles |
|---|---|---|---|
| Reverse | Polymerase Activation and | Ampl | ification |
| Transcription Reaction | cDNA Denaturation | Denaturation | Annealing/Extension |
| 10 min. at 50°C | 1 min. at 95°C | 15 sec. at 95°C | 30 sec. at 60°C |

- 7. We will load the PCR tube onto RT-PCR instrument and allow the RT-qPCR to run.
- 8. E.R. and S.B. will then analyze the RT-PCR products by Melt-Curve Analysis using instrument default setting.

# 4. 4. Sample size:

No sample size could be applied on cell line experiments as we generate millions of naturally randomized cells.

<sup>\*</sup>Qiagen Rotor-Gene®, USA.

### 4. 5. Randomization:

Randomization (with sequence generation and allocation concealment mechanism) is not applied on cell line experiments, as we generate millions of naturally randomized cells, where the amount of cells in each plate will be standardized and each of the 96-well plates will contain the same number of cells (about 25,000-30,000 cells/well).

## 4. 6. Blinding and assessment:

Blinding is not applied on cell line experiments.

### 4. 7. Statistical methodology:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages.

## 5. Results:

## 5. 1. Outcome(s) (O):

- **Primary O:** Apoptosis (Gene expression of Caspase 3).
- > Secondary O: Cytotoxicity/Cell viability.

### 5. 2. Testing the samples:

- 1) After treatment incubation period, E.R. and S.B. will measure the color intensity to estimate cell viability using an ELISA Reader.
- 2) After treatment incubation period, E.R. and S.B. will detect the fold-changes of Caspase 3 gene expression to estimate apoptosis using Rotor-Gene RT-PCR System.

### 6. Protocol amendments:

Any adjustments to the protocol which might affect the conduct of the study, patient's potential benefit or might impact patient safety, including any change in the design of the study, study objectives, methodology, sample sizes, or significant modification in the administrative aspects will require amendment to the protocol formally. Such amendments should be agreed upon by the Council of Oral & Maxillofacial Pathology department.

## 7. Search strategy:

### 7. 1. The PRISMA Statement

### 7. 1. 1. Structured summary:

*Objective:* To estimate the inhibitory effect of luteolin and nano-luteolin as a promoter of cancer cell death in tongue squamous cell carcinoma.

**Data Sources:** In vitro and in vivo articles using PubMed and Cochrane databases. An additional study was identified by contacting the Egyptian Universities Libraries Consortium website (<a href="www.eulc.edu.eg">www.eulc.edu.eg</a>). Search terms included OSCC, TSCC, HNSCC, luteolin and nano-luteolin.

**Study Selection:** Only in vivo and in vitro studies of luteolin (luteolin 5,7,3',4'-tetrahydroxy-flavone) activity regarding apoptosis, cytotoxicity/cell viability on cell lines of oral squamous cell carcinoma (OSCC), tongue squamous cell carcinoma (TSCC) or head and neck squamous cell carcinoma (HNSCC) were included.

**Data Extraction:** Extraction of articles by the author using predefined data fields.

Data Synthesis: Out of all pooled analyses three articles met the inclusion criteria. All trials used luteolin. Apoptosis, cytotoxicity/cell viability were observed to be increased with different doses of luteolin (10 μM for 12 hours) (20-100 μM for 24, 48, 72 hours) (50 μM for 12, 24 hours), separately. Luteolin of 10 μM selectively decreased cell viability and

increased cytotoxicity and apoptosis on tongue squamous cell carcinoma cell line (SCC-25) while increased cell viability on human keratinocyte-derived cell line (HaCaT) versus standard-of-care. When luteolin was used in a dose-dependent and time-dependent pattern the apoptotic cells increased (71%) meanwhile the cell viability decreased (29%) and induced apoptosis selectively on tongue squamous cell carcinoma cell line (SCC-4) and oral cancer cell line (OC-2) versus control. Application of 50 MM of luteolin increased apoptosis of laryngeal HNSCC cell line (Hep-2 cells) versus control.

**Limitations:** Data of results of the included studies is insufficient.

Conclusions: Luteolin between 10 to 100 MM appears to decrease viability and increase cytotoxicity and apoptosis selectively to OSCC, TSCC and HNSCC cell lines.

### 7. 1. 2. Eligibility criteria:

#### 7. 1. 2. 1. Inclusion criteria:

- > Squamous cell carcinoma cell lines (OSCC, TSCC and HNSCC).
- Luteolin 5,7,3',4'-tetrahydroxy-flavone (MeSH term).
- > Application of luteolin as a chemotherapeutic drug.
- ➤ Detection of luteolin activity in apoptosis or cytotoxicity/cell viability.

#### 7. 1. 2. 2. Exclusion criteria:

- Any cancer cell line other than OSCC, TSCC and HNSCC cell lines.
- Luteolin glycosides.
- ➤ Any use of luteolin other than chemotherapy.
- ➤ Detection of luteolin activities other than apoptosis or cytotoxicity/cell viability.

### 7. 1. 2. 3. Report characteristics:

- ➤ No year limitation.
- ➤ No language limitation.

#### 7. 1. 3. Information sources:

Studies were identified by searching electronic databases and scanning reference lists of articles. No limits were applied for language or date of search. This search was first started on 6 May 2017 applied to PubMed and Cochrane electronic databases. The last search was run on 15 June 2017. In addition, the hand search was done through: searching in the department of oral and maxillofacial pathology of Cairo University, checking reference lists of the included articles, searching in the Egyptian Universities Libraries Consortium website <a href="https://www.eulc.edu.eg">www.eulc.edu.eg</a> as well as contacting the authors of the included articles to acquire missing results and there is no reply till now. A limited update literature search was performed from the date of inception till now.

### 7. 1. 4. Synonyms of PICO items:

The following search terms and synonyms were used to search all databases:

| PICO items | Synonyms |
|---|---|
| Fongue squamous cell carcinoma cell line | Tongue squamous cell carcinom* |
| | Tongue squamous cell tumour* |
| | Tongue squamous cell tumor* |
| | Tongue squamous cell neoplasm* |
| | Tongue squamous cell malignan* |
| | Tongue squamous cell cancer* |
| | TSCC |
| | Tongue SCC |
| | Oral tongue squamous cell carcinom* |
| | Oral squamous cell carcinom* |
| | Oral squamous cell tumour* |
| | Oral squamous cell tumor* |
| | Oral squamous cell neoplasm* |
| | Oral squamous cell malignan* |
| | Oral squamous cell cancer* |

| Oral cavity squamous cell carcinom* |
|---------------------------------------|
| OSCC |
| OSCC cell |
| OSCC cell line |
| OSCC cancer |
| Head and neck squamous cell carcinom* |
| Head and neck squamous cell tumour* |
| Head and neck squamous cell tumor* |
| Head and neck squamous cell neoplasm* |
| Head and neck squamous cell malignan* |
| Head and neck squamous cell cancer* |
| HNSCC |
| SCCHN |
| Luteolin |
| Nano-luteolin |
| Nano luteolin |
| Nanoluteolin |
| Luteolin nanoparticles |
| Luteolin nanotechnology |

## 7. 1. 5. **Databases**:

Search Strategy in PubMed and Cochrane, was run on 6 May 2017 till now:

| | Index Term | PubMed | Cochrane |
|-----|-------------------------------------|--------|----------|
| #1 | "Tongue Neoplasms" [MeSH] | 9190 | 56 |
| #2 | tongue squamous cell carcinom* | 781 | 95 |
| #3 | tongue squamous cell tumour* | 1 | 9 |
| #4 | tongue squamous cell tumor* | 7 | 53 |
| #5 | tongue squamous cell neoplasm* | 36 | 54 |
| #6 | tongue squamous cell malignan* | 3 | 5 |
| #7 | tongue squamous cell cancer* | 16 | 70 |
| #8 | tsee | 289 | 6 |
| #9 | tongue scc | 827 | 11 |
| #10 | oral tongue squamous cell carcinom* | 202 | 54 |
| #11 | oral squamous cell carcinom* | 7720 | 816 |
| #12 | oral squamous cell tumour* | 8 | 98 |
| #13 | oral squamous cell tumor* | 42 | 324 |
| #14 | oral squamous cell neoplasm* | 228 | 504 |
| #15 | oral squamous cell malignan* | 10 | 75 |

| #17 oral cavity squamous cell carcinom* | #16 | oral squamous cell cancer* | 112 | 615 |
|---|---|---|---|---|
| #18 osec cell #19 osec cell ine | | 1 | | |
| #19 oscc cell #448 51 #20 oscc cell line 1066 4 #21 oscc cancer 4171 32 #22 head and neck squamous cell carcinom* 7849 1923 #23 head and neck squamous cell tumor* 9 166 #24 head and neck squamous cell tumor* 6 616 #25 head and neck squamous cell tumor* 6 616 #25 head and neck squamous cell malignan* 3 3 84 #27 head and neck squamous cell acancer* 497 1178 #28 hnscc 497 1178 #28 hnscc 5763 303 303 410 or #22 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 20055 2633 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell malignan*) OR (tongue squamous cell carcinom*) OR (tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell cancer*) OR (foral squamous cell cance | | | | |
| #20 oscc cell line #21 oscc cancer #22 head and neck squamous cell carcinom* #349 1923 #23 head and neck squamous cell tumor* 9 166 | | | | |
| #21 oscc cancer #171 32 7849 1923 1924 | | | | |
| #22 head and neck squamous cell tumour* 9 166 #23 head and neck squamous cell tumour* 9 166 #24 head and neck squamous cell tumor* 6 6 616 #25 head and neck squamous cell neoplasm* 377 1029 #26 head and neck squamous cell malignan* 3 84 #27 head and neck squamous cell malignan* 3 84 #28 hnsce 5763 303 #29 sechn 1355 277 #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and ne | | | | |
| #23 head and neck squamous cell tumour* 6 6 616 #24 head and neck squamous cell tumor* 6 6 616 #25 head and neck squamous cell meoplasm* 377 1029 #26 head and neck squamous cell melignan* 3 77 1029 #27 head and neck squamous cell malignan* 3 8 8 4 #27 head and neck squamous cell cancer* 497 1178 #28 hnscc 5763 303 #29 sechn 1355 277 #30 #10 r#20 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumour*) OR (oral squamous cell cancinom*) OR (head and neck squamous cell melplasm*) OR (head and neck squamous cell cancinom*) OR (head and neck squamous cell cancinom*) OR (head and neck squamous cell cancinom*) OR (head and neck squamous cell cancinom*) OR (oral | | | | |
| #24 head and neck squamous cell tumor* #25 head and neck squamous cell neoplasm* #26 head and neck squamous cell malignan* #27 head and neck squamous cell cancer* #27 head and neck squamous cell cancer* #28 hnscc #29 scchn #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumor*) OR (tongue squamous cell tumor*) OR (tongue squamous cell tumor*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell malignan*) OR (oral squamous cell cancer*) OR (osc cancer) OR (head and neck squamous cell neoplasm*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell carcinom*) OR (oral squamous cell cancer*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell carcinom*) OR (oral squamous cell carci | | | | |
| #25 head and neck squamous cell malignan* #26 head and neck squamous cell malignan* #27 head and neck squamous cell cancer* #28 hnscc #29 scchn #30 #10 #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (osec cancer) OR (head and neck squamous cell carcinom*) OR (osec cancer) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell carcinom*) OR (osec cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell malignan*) OR (oral squamous cell carcinom*) OR (oral | | 1 | | |
| #26 head and neck squamous cell malignan* #27 head and neck squamous cell cancer* #28 hnscc #29 sechn #30 #10 r#2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #20 or #21 or #22 or #23 or #24 #30 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 #30 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumorb) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tsce) OR (tongue sce) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell tumorb) OR (oral squamous cell neoplasm*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (osce cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumorb) OR (head and neck squamous cell tumorb) OR (head and neck squamous cell neoplasm*) OR (head and neck squamous cell malignan*) OR (tongue squamous cell tumourb) OR (tongue squamous cell tumorb) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell carcinomb) OR (tongue squamous cell carcinomb) OR (tongue squamous cell carcinomb) OR (tongue squ | | 1 | | |
| #27 head and neck squamous cell cancer* #28 hnscc #29 scchn #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tongue squamous cell malignan*) OR (oral squamous cell cancer*) OR (oral squamous cell carcinom*) OR (oral squamous cell cancer*) OR (oral squamous cell cancer*) OR (oral squamous cell cancer*) OR (oral squamous cell cancer*) OR (oral squamous cell cancer*) OR (osec cancer) OR (head and neck squamous cell cancer*) OR (oral squamous cell cancer*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell cancer*) OR (head and neck squamous c | | 1 1 | | |
| #28 hnscc 5763 303 #29 sechn 1355 277 #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 20055 2633 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (toral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell malignan*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oscc cancer) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell m | | ı e | | |
| #29 scchn #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell tumor*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell carcinom*) OR (osec cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell carcinom*) OR (bead and neck squamous cell carcinom*) OR (bead and neck squamous cell carcinom*) OR (bead and neck squamous cell carcinom*) OR (tongue squamous cell tumor*) OR (tongue squamous cell malignan*) OR (tongue squamous cell carcinom*) OR (tongue squamous cell carcinom*) OR (tongue squamous cell carcinom*) OR (tongue squamous cell carcinom*) OR (tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (bead and neck squamous cell carcinom*) OR (bead and neck squamous cell carcinom*) OR (bead and neck squamous cell carcinom*) OR (bead and neck squamous cell carcin | | | | |
| #30 #1 or #2 or #3 or #4 or #5 or #6 or #7 or #8 or #9 or #10 or #11 or #12 or #13 or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tscc) OR (tongue scc) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oscc oracer*) OR (head and neck squamous cell carcinom*) OR (oscc cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell tumor*) OR (tongue squamous cell malignan*) OR (tongue squamous cell malignan*) OR (tongue squamous cell malignan*) OR (tongue squamous cell malignan*) OR (tongue squamous cell malignan*) OR (tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell carcinom*) OR (or | | | | |
| or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 or #25 or #26 or #27 or #28 or #29 (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumour*) OR (tongue squamous cell cancer*) OR (tscc) OR (tongue scc) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oscc cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell malignan*) OR (tongue squamous cell tumor*) OR (tongue squamous cell tumor*) OR (tongue squamous cell tumor*) OR (tongue squamous cell tumor*) OR (tongue squamous cell cancer*) OR (tongue squamous cell cancer*) OR (tongue squamous cell cancer*) OR (tongue squamous cell cancer*) OR (tongue squamous cell cancer*) OR (oral cavity squamous cell cancers*) OR (oral squamous cell cancers*) OR (oral cavity squamous cell cancers*) OR (oral squamous cell cancers*) OR (oral cavity squamous cell cancers*) OR (oral squamous cell cancers*) OR (oral cavity squamous cell cancers*) OR (oral squamous cell cancers*) OR (oral cavity squamous cell cancers*) OR (head and neck squamous cell cancers*) OR (head and | | | | |
| (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tsec) OR (tongue sec) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell neoplasm*) OR (oral squamous cell malignan*) OR (oral squamous cell neoplasm*) OR (oral squamous cell carcinom*) OR (oscc cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell cancer*) OR (hnscc) OR (scchn) #31 #1 or #30 | #30 | or #14 or #15 or #16 or #17 or #18 or #19 or #20 or #21 or #22 or #23 or #24 | 20033 | 2033 |
| ("Tongue Neoplasms" [Mesh]) OR (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tongue scc) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumour*) OR (oral squamous cell tumor*) OR (oral squamous cell neoplasm*) OR (oral squamous cell malignan*) OR (oral squamous cell cancer*) OR (oral cavity squamous cell carcinom*) OR (oscc) OR (oscc cell) OR (oscc cell line) OR (oscc cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell neoplasm*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell cancer*) OR (head and neck squamous cell cancer*) OR (head ond | | (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tscc) OR (tongue scc) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell tumor*) OR (oral squamous cell neoplasm*) OR (oral squamous cell malignan*) OR (oral squamous cell cancer*) OR (oral cavity squamous cell carcinom*) OR (oscc) OR (oscc cell) OR (oscc cell line) OR (oscc cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell cancer*) OR (hnscc) OR | | |
| #32 "Luteolin"[Mesh] 1263 2 | #31 | ("Tongue Neoplasms" [Mesh]) OR (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tscc) OR (tongue scc) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell neoplasm*) OR (oral squamous cell malignan*) OR (oral squamous cell cancer*) OR (oral cavity squamous cell carcinom*) OR (oscc) OR (oscc cell) OR (oscc cell line) OR (oscc cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumor*) OR (head and neck squamous cell neoplasm*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell | 27867<br>1263 | 2660 |

| #33 | Luteolin | 3224 | 18 |
|---|---|---|---|
| #34 | #32 or #33 | 3224 | 18 |
| | ("Luteolin"[Mesh]) or (Luteolin) | _ | |
| #35 | nano-luteolin | 1 | 0 |
| #36 | nano luteolin | 11 | 0 |
| #37 | Nanoluteolin | 0 | 0 |
| #38 | luteolin nanoparticles | 19 | 0 |
| #39 | luteolin nanotechnology<br>#35 or #36 or #37 or #38 or #39 | 8<br>31 | 0 |
| #40 | #33 01 #30 01 #37 01 #38 01 #39 | 31 | U |
| | (nano-luteolin) OR (nano luteolin) OR (nanoluteolin) OR (luteolin | | |
| | nanoparticles) OR (luteolin nanotechnology) | | |
| #41 | #34 and #40 | 31 | 0 |
| | | | • |
| | ("Luteolin" [Mesh]) OR (luteolin) AND (nano-luteolin) OR (nano luteolin) | | |
| | OR (nanoluteolin) OR (luteolin nanoparticles) OR (luteolin nanotechnology) | | |
| #42 | #31 and #34 | 6 | 0 |
| | ("Tongue Neoplasms" [Mesh]) OR (tongue squamous cell carcinom*) OR | | |
| | (tongue squamous cell tumour*) OR (tongue squamous cell tumor*) OR | | |
| | (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR | | |
| | (tongue squamous cell cancer*) OR (tscc) OR (tongue scc) OR (oral tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral | | |
| | squamous cell tumour*) OR (oral squamous cell tumor*) OR (oral squamous | | |
| | cell neoplasm*) OR (oral squamous cell malignan*) OR (oral squamous cell | | |
| | cancer*) OR (oral cavity squamous cell carcinom*) OR (osco) OR (osco cell) | | |
| | OR (oscc cell line) OR (oscc cancer) OR (head and neck squamous cell | | |
| | carcinom*) OR (head and neck squamous cell tumour*) OR (head and neck | | |
| | squamous cell tumor*) OR (head and neck squamous cell neoplasm*) OR | | |
| | (head and neck squamous cell malignan*) OR (head and neck squamous cell | | |
| | cancer*) OR (hnscc) OR (scchn) AND ("Luteolin"[Mesh]) or (Luteolin) | | |
| #43 | #31 and #40 | 1 | 0 |
| 1 | (UT) N. 1 U FN 1N OP ( | | |
| | ("Tongue Neoplasms" [Mesh]) OR (tongue squamous cell carcinom*) OR | | |
| | (tongue squamous cell tumour*) OR (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR | | |
| | (tongue squamous cell cancer*) OR (tscc) OR (tongue scc) OR (oral tongue | | |
| | squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral | | |
| | squamous cell tumour*) OR (oral squamous cell tumor*) OR (oral squamous | | |
| | cell neoplasm*) OR (oral squamous cell malignan*) OR (oral squamous cell | | |
| | cancer*) OR (oral cavity squamous cell carcinom*) OR (oscc) OR (oscc cell) | | |
| | OR (oscc cell line) OR (oscc cancer) OR (head and neck squamous cell | | |
| | carcinom*) OR (head and neck squamous cell tumour*) OR (head and neck | | |
| | squamous cell tumor*) OR (head and neck squamous cell neoplasm*) OR | | |
| İ | (head and neck squamous cell malignan*) OR (head and neck squamous cell | | |
| İ | cancer*) OR (hnscc) OR (scchn) AND (nano-luteolin) OR (nano luteolin) OR | | |
| | (nanoluteolin) OR (luteolin nanoparticles) OR (luteolin nanotechnology) | | |

| #44 | #31 and #34 and #40 | 1 | 0 |
|---|---|---|---|
| | ("Tongue Neoplasms" [Mesh]) OR (tongue squamous cell carcinom*) OR (tongue squamous cell tumour*) OR (tongue squamous cell tumor*) OR (tongue squamous cell neoplasm*) OR (tongue squamous cell malignan*) OR (tongue squamous cell cancer*) OR (tongue squamous cell malignan*) OR (tongue squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell carcinom*) OR (oral squamous cell tumor*) OR (oral squamous cell neoplasm*) OR (oral squamous cell malignan*) OR (oral squamous cell cancer*) OR (oral cavity squamous cell carcinom*) OR (oscc) OR (oscc cell) OR (oscc cell line) OR (oscc cancer) OR (head and neck squamous cell carcinom*) OR (head and neck squamous cell tumour*) OR (head and neck squamous cell neoplasm*) OR (head and neck squamous cell malignan*) OR (head and neck squamous cell cancer*) OR (hnscc) OR (scchn) AND ("Luteolin"[Mesh]) or (Luteolin) AND (nano-luteolin) OR (nano luteolin) OR (nanoluteolin) OR (luteolin nanoparticles) OR (luteolin nanotechnology) | | |

### 7. 1. 6. Study selection:

The search started with 7 articles. The retrieved records were screened on the basis of title and abstract and sequentially two out of them were excluded according to the exclusion criteria. (The used cell lines were human breast cancer adenocarcinoma, human colon colorectal carcinoma and human hepatic carcinoma cell lines, not OSCC, TSCC or HNSCC cell lines (n=1), and luteolin glycosides were used with different molecular formula than luteolin 5,7,3',4'-tetrahydroxy-flavone (n=1)). Manuscript review and application of inclusion criteria of the remaining five articles with full text publication were done. This resulted in Reasonable exclusion of two additional articles. (Luteolin was used in chemoprevention not as a chemotherapeutic drug (n=1), and luteolin was used to detect different outcomes other than apoptosis or cytotoxicity/cell viability (n=1)). The three remaining full-text articles met the eligibility criteria and included to extract data out of them. For note, each stage of these steps was carried out only by the author.

#### PRISMA flow diagram of study selection:



### 7. 1. 7. Data collection process:

Information was extracted from each included study and refined accordingly. The authors of the included studies were contacted for information that is unclearly reported. However, there is no answer till now.

#### 7. 1. 8. Data items:

Information were extracted from each included study on: (1) characteristics of trial population (including number of groups), and the trial's inclusion and exclusion criteria; (2) type of intervention (including type, dose, duration versus control, standard-of-care or versus no treatment), (3) type of outcome measure (including apoptosis and cytotoxicity/cell viability).

# 7. 2. Summary of finding tables (SOFT):

# 7. 2. 1. Demographics of included studies:

| No.<br>of<br>study | Study 1st<br>Author<br>(Year/<br>country) | Name of journal | Title of the study | Type of samples | Control | Type of study | Source |
|---|---|---|---|---|---|---|---|
| 1 | K.C.<br>Tjioe,<br>France<br>2016 | Nutrition And<br>Cancer | Luteolin Impacts on the DNA Damage Pathway in Oral Squamous Cell Carcinoma | 1- Tongue<br>squamous cell<br>carcinoma cell<br>line (SCC-25<br>cells)<br>2- Human<br>keratinocyte-<br>derived cell<br>line (HaCaT) | DMSO | In vitro | PubMed |
| 2 | S. F.<br>Yang,<br>Taiwan<br>2008 | J Dent Res | Luteolin Induces Apoptosis in Oral Squamous Cancer Cells | 1- Tongue<br>squamous cell<br>carcinoma cell<br>line (SCC-4<br>cells)<br>2-Oral cancer<br>cell line (OC-<br>2 cells) | DMSO | In vitro<br>and In<br>vivo<br>(Animal) | PubMed |
| 3 | H.<br>Zhang,<br>China<br>2014 | Eur Arch<br>Otorhinolaryngol | Luteolin induces apoptosis by activating Fas signaling pathway at the receptor level in laryngeal squamous cell line Hep.2 cells | - Laryngeal<br>HNSCC cell<br>line (Hep-2<br>cells) | DMSO | In vitro | PubMed |

### 7. 2. 2. Material and Methods:

| | | 0 | | | | | МТ | T as | say | Cr | ystal | viole | t staining | | | | Western | blot | | D | API | staining | I | Flow | cytom | etric analysis | RT-PCR | | | R |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. of study | Cell line types | Culture media | Drug | Groups | Control | Standard-of- | Dose | Duration | Material | Control<br>Groups | Dose | Duration | Material | Control | Dose | Duration | Antibodies | Material | Control | Dose | Duration | Material | Dose | Duration | Protein | Material | Housekeeping | Primer | Antibodies | Material |
| 1 | 1-SCC-25 2-HaCaT | DMEM/F12<br>10% FBS<br>1% penicillin<br>and<br>streptomycin<br>400ng/ml of<br>hydro-<br>cortisone<br>15mM N-2<br>HEPES | Luteolin | NA | | CP / | 5,10,20 MM 5,10 MM 10 MM | 72, 24, 48, 72 h | Colorimetric assay 1-(4,5-dimethyl-thiazol-2-yl)-3 5-diphenyl formazan Thiazolyl blue formazan 25ml of MTT reagent | 6-well plate (25,000 cells/well) | 10 mM | 72 h | Glutaral-dehyde 2%, PBS, Crystal violet 0.05%, Acetic acid 1% | Nil | 10 MM | 30 min | p-JNK p-EGFR p-AKT p- p38 p-ERK1/2<br>p-ATM p-ATR p- H2AX p-CHK2 p-<br>BRCA1 ERK1/2 JNK1/2 ERK2 CHK2 | TNT buffer,<br>MicroBCA kit<br>(30 mg/well)<br>NuPAGE<br>electrophoresis<br>Nitrocellulose<br>membranes | | | No | t used | | | Not | used | | | Not used | 1 |
| 2 | 1-SCC-4 2-OC-2 | DMEM/F12<br>10% FBS<br>1% penicillin<br>and<br>streptomycin<br>400ng/ml of<br>hydro-<br>cortisone<br>2 mM<br>glutamine | Luteolin | 24-well plate | DMSO | P | 5, 10 MM 0-100 MM 0.3 | 24, 48, 72 h 24, 48, | 0.5 mg/mL<br>MTT<br>reagent, Blue<br>formazan<br>crystals | | N | Not us | sed | ß-actin | 0-100 MM | NA | Bcl-2 Bax Caspase9 Caspase 3 PARP | NA | Nii | 0-100 mM | 48 h | 4',6-<br>Diamidino<br>-2-<br>phenylindol<br>e (DAPI)<br>(1 mg/ml) | MH 001-0 | 24 h | NA | NA | | | Not used | i |
| 3 | Hep-2 cells | DMEM/F12<br>penicillin<br>and<br>streptomycin | Luteolin | NA | DMSO | No | 20-100 MM | NA | 3-(4,5-dimethyl-thiazol-2-yl)-2,5-diphenyl tetrazolium bromide (MTT) | | Ŋ | Vot us | sed | β-actin | 0.30.50 MM | 6, 12, 24 h | anti-c-FLIPS/L anti-Fas<br>per-oxidase-conjugated goat<br>anti-rabbit 2ry antibody | SDS/PAGE<br>(12 % w/v)<br>Nitrocellulose<br>membranes<br>non-fat milk<br>(5 %)<br>TBST | DMSO | 0.30.50 MM | 24 h | 4',6-<br>Diamidino-<br>2-<br>phenylindol<br>e(DAPI) | 50 uM | 6, 12, 24 h | Caspase3, Caspase 8, Caspase 9 | Annexin V-FITC Apoptosis Detection Kit Becton-Dickinson CELL Quest software | β-actin | 8-12 | c-FLIP Fas IgG peroxidase-conjugated 2ry antibody | Aliquots<br>of PCR<br>products<br>agarose<br>gel (1.5<br>%)<br>electropho<br>resis<br>ethidium<br>bromide |

### 7. 2. 3. Results:

| | | Apoptosis | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. of the study | Drug | | 1 | Antibodies | | | | Duratio | Dose | Effect | | |
| | | p-JNK | Caspase-3 | Caspase-9 | cFLIP <sub>L</sub> | 6 h | 12 h | 24 h | 48 h | 72 h | Dose | Direct |
| 1 | Luteolin | p-JNK | _ | - | - | _ | _ | _ | _ | 72 h | 10 μΜ | 0.34 fold |
| 2 | Luteolin | _ | Caspase-3 | - | - | ı | ı | _ | 48 h | ı | 60-100 μΜ | 32 kDa |
| 2 | Luteolin | _ | _ | Caspase-9 | _ | 1 | - | _ | 48 h | - | 60-100 μΜ | 47 kDa |
| | Luteolin | _ | _ | - | $cFLIP_L$ | 6 h | _ | _ | _ | _ | 30 μΜ | 0.65 fold |
| | Luteolin | _ | _ | - | $cFLIP_L$ | 6 h | - | _ | - | - | 50 μΜ | 0.40 fold |
| | Luteolin | _ | _ | _ | cFLIP <sub>L</sub> | ı | 12 h | _ | _ | _ | 30 μΜ | 0.38 fold |
| 3 | Luteolin | _ | _ | - | $cFLIP_L$ | - | 12 h | _ | - | - | 50 μM | 0.19 fold |
| | Luteolin | _ | _ | - | cFLIP <sub>L</sub> | _ | _ | 24 h | _ | _ | 30 μΜ | 0.15 fold |
| | Luteolin | _ | _ | _ | cFLIP <sub>L</sub> | - | _ | 24 h | _ | _ | 50 μΜ | 0.13 fold |

| | | Cytotoxicity/Cell viability (%) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| No. of the study | Drug | | | Dose | Effect | | | |
| | | 6 h | 12 h | 24 h | 48 h | 72 h | | |
| 1 | Luteolin | _ | _ | _ | _ | 72 h | 20 μΜ | 83.33% |
| | Luteolin | - | _ | 24 h | _ | _ | 60 μΜ | 0.12 *104% |
| | Luteolin | _ | _ | 24 h | _ | _ | 80 μΜ | 0.15*10 <sup>4</sup> % |
| | Luteolin | _ | _ | 24 h | _ | _ | 100 μΜ | 0.17*10 <sup>4</sup> % |
| | Luteolin | _ | - | I | 48 h | _ | 60 μΜ | 0.63*10 <sup>4</sup> % |
| 2 | Luteolin | _ | _ | _ | 48 h | _ | 80 μΜ | 1.08*10 <sup>4</sup> % |
| | Luteolin | _ | _ | - | 48 h | | 100 μΜ | 1.60*10 <sup>4</sup> % |
| | Luteolin | _ | _ | _ | _ | 72 h | 60 μΜ | 1.17*10 <sup>4</sup> % |
| | Luteolin | _ | _ | _ | _ | 72 h | 80 μΜ | 1.75*10 <sup>4</sup> % |
| | Luteolin | _ | - | - | - | 72 h | 100 μΜ | 2.35*10 <sup>4</sup> % |
| | Luteolin | 6 h | - | I | _ | _ | 50 μΜ | 4.33 % |
| 3 | Luteolin | _ | 12 h | _ | _ | _ | 50 μΜ | 4.66 % |
| | Luteolin | _ | - | 24 h | _ | _ | 50 μΜ | 16.00 % |

## 7. 2. 4. Table of excluded studies:

| No. of study | Study 1st Author (Country, Year) | Journal | Title of study | Reason of exclusions | Source |
|---|---|---|---|---|---|
| 1 | L. Gohar,<br>Egypt 2016 | International Journal of Pharmacognosy and Phytochemistry | Phytochemical and<br>Biological Studies of<br>Certain Plants<br>Possessing Cytotoxic<br>Activity | Human breast cancer<br>adenocarcinoma, Human<br>colon colorectal carcinoma<br>and Human hepatic<br>carcinoma cell lines. <b>NOT</b><br>OSCC, TSCC or HNSCC<br>cell lines | www.eulc.edu.eg |
| 2 | T. Matsuta,<br>Japan 2011 | In Vivo | Biological Activity of<br>Luteolin Glycosides<br>and Tricin from Sasa<br>senanensis Rehder | Application of Luteolin glycosides. <b>NOT</b> the molecular formula Luteolin 5,7,3',4'-tetrahydroxy-flavone | PubMed |
| 3 | D. Majumdar,<br>USA 2014 | Cancer Prev<br>Res | Luteolin nanoparticle in chemoprevention – in vitro and in vivo anticancer activity | Application of luteolin in chemopevention. <b>NOT</b> as a chemotherapeutic drug | PubMed |
| 4 | R. B. Selvi,<br>India 2015 | Oncotarget | Inhibition of p300 lysine acetyltransferase activity by luteolin reduces tumor growth in head and neck squamous cell carcinoma (HNSCC) xenograft mouse model | Detection of p300<br>KAT/p300 acetyl-<br>transferase and cancer<br>progression activity. <b>NOT</b><br>detecting apoptosis or<br>cytotoxicity/cell viability. | PubMed |

### 8. References:

- 1. WHO | Cancer. WHO [Internet]. 2017 [cited 2017 Apr 13]; Available from: http://www.who.int/mediacentre/factsheets/fs297/en/#.WO8mcUySM2c.men deley&title=Cancer&description=Cancer is a generic term for a large group of diseases that can affect any part of the body.
- 2. Warnakulasuriya S. Global epidemiology of oral and oropharyngeal cancer. Oral Oncol [Internet]. 2009;45(4–5):309–16. Available from: http://dx.doi.org/10.1016/j.oraloncology.2008.06.002
- 3. Aruna DS, Prasad KV V, Shavi GR, Ariga J, Rajesh G, Krishna M. Retrospective study on risk habits among oral cancer patients in karnataka cancer therapy and research institute, hubli, India. Asian Pacific J Cancer Prev. 2011;12(6):1561–6.
- 4. Huang S-H, O'sullivan B. Oral cancer: Current role of radiotherapy and chemotherapy. Med Oral Patol Oral Cir Bucal Mar Mar Med Oral S L CIF B Med Oral Patol Oral Cir Bucal Mar [Internet]. 2013;1181818(12):233–40. Available from: http://www.medicinaoral.com/medoralfree01/v18i2/medoralv18i2p233.pdf% 5Cnhttp://www.medicinaoral.com/:10.4317/medoral.18772%5Cnhttp://dx.doi.org/doi:10.4317/medoral.18772
- 5. Neville BW. Oral and maxillofacial pathology [Internet]. 3rd ed. Elsevier; 2009. 984 p. Available from: https://evolve.elsevier.com/cs/product/9781416034353?
- 6. Liu H, Dong Y, Gao Y, Du Z, Wang Y, Cheng P, et al. The fascinating effects of baicalein on cancer: A review. Int J Mol Sci. 2016;17(10).
- 7. Romano B, Pagano E, Montanaro V, Fortunato AL, Milic N, Borrelli F. Novel insights into the pharmacology of flavonoids. Phyther Res. 2013;27(11):1588–96.
- 8. Russo M, Spagnuolo C, Tedesco I, Russo GL. Phytochemicals in cancer prevention and therapy: Truth or dare? Toxins (Basel). 2010;2(4):517–51.

- 9. Chen Z, Kong S, Song F, Li L, Jiang H. Pharmacokinetic study of luteolin, apigenin, chrysoeriol and diosmetin after oral administration of Flos Chrysanthemi extract in rats. Fitoterapia [Internet]. 2012 [cited 2017 Apr 1];83(8):1616–22. Available from: http://www.sciencedirect.com/science/article/pii/S0367326X12002584
- 10. Kim YA, Yu JG, Lee KW, Lee HJ. Luteolin suppresses UVB-induced photoageing by targeting. 2013;17(5):672–80.
- 11. Miean KH, Mohamed S. Flavonoid (Myricetin, Quercetin, Kaempferol, Luteolin, and Apigenin) Content of Edible Tropical Plants. J Agric Food Chem [Internet]. 2001 Jun 1;49(6):3106–12. Available from: http://dx.doi.org/10.1021/jf000892m
- 12. Sun T, Xu Z, Wu CT, Janes M, Prinyawiwatkul W, No HK. Antioxidant activities of different colored sweet bell peppers (Capsicum annuum L.). J Food Sci. 2007;72(2):98–102.
- 13. Seelinger G, Merfort I, Wölfle U, Schempp CM. Anti-carcinogenic Effects of the Flavonoid Luteolin. 2008;2628–51.
- 14. Majumdar D, Jung KH, Zhang H, Nannapaneni S, Wang X, Ruhul Amin ARM, et al. Luteolin nanoparticle in chemoprevention: In vitro and in vivo anticancer activity. Cancer Prev Res. 2014;7(1):65–73.
- 15. Ding S, Hu A, Hu Y, Ma J, Weng P, Dai J. Anti-hepatoma cells function of luteolin through inducing apoptosis and cell cycle arrest. Tumour Biol J Int Soc Oncodevelopmental Biol Med [Internet]. 2014;35(4):3053–60. Available from: http://search.ebscohost.com/login.aspx?direct=true&db=cmedm&AN=24287 949&site=ehost-live
- 16. Calixto G, Fonseca-Santos B, Chorilli M, Bernegossi J. Nanotechnology-based drug delivery systems for treatment of oral cancer: a review. Int J Nanomedicine [Internet]. 2014;9(1):3719. Available from: http://www.dovepress.com/nanotechnology-based-drug-delivery-systems-for-treatment-of-oral-cance-peer-reviewed-article-IJN

- 17. Chalovich JM, Eisenberg E. NIH Public Access. Biophys Chem. 2005;257(5):2432–7.
- 18. Takahashi Y, Hamada J, Murakawa K, Takada M, Tada M, Nogami I, et al. Expression profiles of 39 HOX genes in normal human adult organs and anaplastic thyroid cancer cell lines by quantitative real-time RT-PCR system. 2004;293:144–53.
- 19. Journal E. Comparison Of The Sulforhodamine-B Protein And Tetrazolium (MTT) Assays For Invitro Chemosensitivity Testing. 1991;5379(February).